CLINICAL TRIAL: NCT01367132
Title: Assessment of the Number of Umbilical Cord Vessels at the Time of Nuchal Translucency Screening
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MedStar 2010-450
Record Dates: First submitted 2011-06-01; First posted 2011-06-06 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Umbilical Cord
Keywords: ultrasound; first trimester; umbilical cord

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Doppler ultrasound — Ultrasound using Doppler mode to detect blood flow in umbilical cord vasculature and determine the number of vessels present

SUMMARY:
The primary objective of this study is to determine the detection rate of two- or three-vessel umbilical cord at the time of nuchal translucency screening between 11 and 13 6/7 weeks gestation.

Hypothesis: Detection rate of the number of vessels during first trimester will be as accurate as the detection of vessels during the second trimester.

ELIGIBILITY:
Inclusion Criteria:

* Singleton or multiple-gestation pregnancies in patients presenting for NT screening between 11 and 13 6/7 weeks gestation and CRL between 45-84mm as determined at the time of the ultrasound
* Age 18 and older

Exclusion Criteria:

* Patients who are incapable of informed consent or minors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing nuchal transluscency screening during 11-13+6 weeks gestation, followed by anatomy scan at 18-24 weeks gestation.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Detection of the number of vessels in the umbilical cord between 11 and 13 6/7 weeks. | 11-13+6 weeks
Detection of the number of vessels in the umbilical cord between 18 and 23 6/7 weeks. | 18 - 23 6/7 weeks

SECONDARY OUTCOMES:
Sensitivity and specificity of transabdominal sonography at detecting vasculature of the cord between 11 and 13 6/7 weeks. | 11-13+6 weeks gestational age
Sensitivity and specificity of transabdominal sonography at detecting vasculature of the cord during the second trimester. | 18-24 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Rita W Driggers, MD, Principal Investigator — Washington Hospital Center, MedStar Health
Locations (2):
- United States (2):
  - Georgetown University Hospital, MedStar Health, Washington D.C., District of Columbia
  - Washington Hospital Center, MedStar Health, Washington D.C., District of Columbia

REFERENCES:
- [Background] Cuckle H, Nanchahal K, Wald N. Birth prevalence of Down's syndrome in England and Wales. Prenat Diagn. 1991 Jan;11(1):29-34. doi: 10.1002/pd.1970110106. PMID 1827525
- [Background] ACOG Committee on Practice Bulletins. ACOG Practice Bulletin No. 77: screening for fetal chromosomal abnormalities. Obstet Gynecol. 2007 Jan;109(1):217-27. doi: 10.1097/00006250-200701000-00054. PMID 17197615
- [Background] Souka AP, Nicolaides KH. Diagnosis of fetal abnormalities at the 10-14-week scan. Ultrasound Obstet Gynecol. 1997 Dec;10(6):429-42. doi: 10.1046/j.1469-0705.1997.10060429.x. No abstract available. PMID 9476332
- [Background] Dugoff L. Ultrasound diagnosis of structural abnormalities in the first trimester. Prenat Diagn. 2002 Apr;22(4):316-20. doi: 10.1002/pd.309. PMID 11981912
- [Background] Whitlow BJ, Chatzipapas IK, Lazanakis ML, Kadir RA, Economides DL. The value of sonography in early pregnancy for the detection of fetal abnormalities in an unselected population. Br J Obstet Gynaecol. 1999 Sep;106(9):929-36. doi: 10.1111/j.1471-0528.1999.tb08432.x. PMID 10492104
- [Background] Economides DL, Whitlow BJ, Braithwaite JM. Ultrasonography in the detection of fetal anomalies in early pregnancy. Br J Obstet Gynaecol. 1999 Jun;106(6):516-23. doi: 10.1111/j.1471-0528.1999.tb08317.x. No abstract available. PMID 10426606
- [Background] Becker R, Wegner RD. Detailed screening for fetal anomalies and cardiac defects at the 11-13-week scan. Ultrasound Obstet Gynecol. 2006 Jun;27(6):613-8. doi: 10.1002/uog.2709. PMID 16570262
- [Background] Abu-Rustum RS, Daou L, Abu-Rustum SE. Role of ultrasonography in early gestation in the diagnosis of congenital heart defects. J Ultrasound Med. 2010 May;29(5):817-21. doi: 10.7863/jum.2010.29.5.817. PMID 20427794
- [Background] Lombardi CM, Bellotti M, Fesslova V, Cappellini A. Fetal echocardiography at the time of the nuchal translucency scan. Ultrasound Obstet Gynecol. 2007 Mar;29(3):249-57. doi: 10.1002/uog.3948. PMID 17318942
- [Background] Heifetz SA. The umbilical cord: obstetrically important lesions. Clin Obstet Gynecol. 1996 Sep;39(3):571-87. doi: 10.1097/00003081-199609000-00007. No abstract available. PMID 8862884
- [Background] Murphy-Kaulbeck L, Dodds L, Joseph KS, Van den Hof M. Single umbilical artery risk factors and pregnancy outcomes. Obstet Gynecol. 2010 Oct;116(4):843-850. doi: 10.1097/AOG.0b013e3181f0bc08. PMID 20859147
- [Background] Parilla BV, Tamura RK, MacGregor SN, Geibel LJ, Sabbagha RE. The clinical significance of a single umbilical artery as an isolated finding on prenatal ultrasound. Obstet Gynecol. 1995 Apr;85(4):570-2. doi: 10.1016/0029-7844(94)00451-I. PMID 7898835
- [Background] Heifetz SA. Single umbilical artery. A statistical analysis of 237 autopsy cases and review of the literature. Perspect Pediatr Pathol. 1984 Winter;8(4):345-78. PMID 6514541
- [Background] Hill LM, Wibner D, Gonzales P, Chenevey P. Validity of transabdominal sonography in the detection of a two-vessel umbilical cord. Obstet Gynecol. 2001 Nov;98(5 Pt 1):837-42. doi: 10.1016/s0029-7844(01)01572-1. PMID 11704178
- [Background] Rembouskos G, Cicero S, Longo D, Sacchini C, Nicolaides KH. Single umbilical artery at 11-14 weeks' gestation: relation to chromosomal defects. Ultrasound Obstet Gynecol. 2003 Dec;22(6):567-70. doi: 10.1002/uog.901. PMID 14689527
- [Background] Nyberg DA, Mahony BS, Luthy D, Kapur R. Single umbilical artery. Prenatal detection of concurrent anomalies. J Ultrasound Med. 1991 May;10(5):247-53. doi: 10.7863/jum.1991.10.5.247. PMID 2051544
- [Background] Sheiner E, Shoham-Vardi I, Hussey MJ, Pombar X, Strassner HT, Freeman J, Abramowicz JS. First-trimester sonography: is the fetus exposed to high levels of acoustic energy? J Clin Ultrasound. 2007 Jun;35(5):245-9. doi: 10.1002/jcu.20321. PMID 17410588
- [Background] Sheiner E, Shoham-Vardi I, Pombar X, Hussey MJ, Strassner HT, Abramowicz JS. An increased thermal index can be achieved when performing Doppler studies in obstetric sonography. J Ultrasound Med. 2007 Jan;26(1):71-6. doi: 10.7863/jum.2007.26.1.71. PMID 17182711
- [Background] American Institute of Ultrasound in Medicine. AIUM practice guideline for the performance of obstetric ultrasound examinations. J Ultrasound Med. 2010 Jan;29(1):157-66. doi: 10.7863/jum.2010.29.1.157. No abstract available. PMID 20040792
- [Background] Barnett SB, Maulik D; International Perinatal Doppler Society. Guidelines and recommendations for safe use of Doppler ultrasound in perinatal applications. J Matern Fetal Med. 2001 Apr;10(2):75-84. doi: 10.1080/714904312. PMID 11392597